CLINICAL TRIAL: NCT02099760
Title: A Validation Study of the Cepheid Xpert CT/NG for Detecting Chlamydia Trachomatis and Neisseria Gonorrhoeae in Rectal Samples
Brief Title: Cepheid Rectal Sample Validation Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Sharon Hillier, Professor, University of Pittsburgh
Other Study IDs: PRO13100170; 5U01AI068633-04 (NIH)
Record Dates: First submitted 2014-03-12; First posted 2014-03-31 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Gonorrhea; Chlamydia; Trichomonas
Keywords: gonorrhea; chlamydia; trichomonas
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Trichomonas Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Any leftover specimens including genital, rectal, pharyngeal, or urine may be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STD testing (GC/Ct/trich)
  Interventions: Device: STD testing (GC/Ct/trich)

INTERVENTIONS:
Device: STD testing (GC/Ct/trich)
  Other Names: Cepheid Xpert CT/NG

SUMMARY:
The purpose of this study is to validate Xpert CT/NG for the detection of CT and GC in rectal samples as part of the PA DOH and CLIA requirements. The evaluation of samples obtained from the pharynx is exploratory and will provide new information on the frequency of pharyngeal infection due to CT and GC.

A secondary objective will be to evaluate the prevalence of Trichomonas vaginalis in vaginal and rectal samples using both the Xpert system and AC2 to assess whether women positive for this pathogen rectally usually or always have vaginal infection due to this pathogen.

The investigators hypothesis is that real-time PCR (polymerase chain reaction) amplification testing with the Cepheid Xpert CT/NG will have greater sensitivity than culture in detecting Neisseria gonorrhoeae in rectal samples. The investigators also hypothesize that Xpert CT/NG will be equivalent to the Gen-Probe APTIMA Combo2 (AC2) in detecting Chlamydia trachomatis and Neisseria gonorrhoeae in rectal samples.

DETAILED DESCRIPTION:
Because of its high sensitivity and specificity, NAAT testing has largely replaced bacterial culture for the diagnosis of genital CT and GC in both males and females. NAAT assays have the greatest potential for detecting CT and GC in the rectum; however, no NAAT is currently cleared for use with extragenital specimens by the US Food and Drug Administration.

In order to comply with CLIA regulations, laboratories must perform in-house validations to use NAATs with rectal and pharyngeal specimens. There are multiple studies in the literature evaluating NAAT assays in diagnosing CT and GC in rectal and pharyngeal specimens using expanded reference standards, which includes positive culture result and secondary confirmatory NAAT assays. The proposed validation study is intended to provide data to support the use of NAAT for rectal and pharyngeal specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18 and older
2. Women or men who have a history of engaging in receptive anal intercourse
3. Willing to provide written informed consent for participation in this study

Exclusion Criteria:

1. Use of oral antibiotics in the past 7 days
2. Use of rectal douche or other rectal product in the past 24 hours
3. If female, use of a vaginal douche or vaginal product in the past 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects presenting for routine clinical care in an STD Clinic and/or subjects who are aware of the study and meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Rectal Gonorrhea/Chlamydia testing result | approximately 7 days
  Compare the sensitivity and specificity of the Xpert NG to the AC2 and culture in detecting GC in rectal samples Compare the sensitivity and specificity of the Xpert CT to AC2 (and as necessary, for discrepant results, to Aptima CT assay) in detecting CT in rectal samples

SECONDARY OUTCOMES:
pharyngeal GC/Ct result | approximately 7 days
  The evaluation of samples obtained from the pharynx is exploratory and will provide new information on the frequency of pharyngeal infection due to CT and GC.
Trichomonas Testing Results | approximately 7 days
  evaluate the prevalence of Trichomonas vaginalis in vaginal and rectal samples using both the Xpert system and AC2

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hillier, PhD, Principal Investigator — University of Pittsburgh/UPMC
Locations (2):
- United States (2):
  - Allegheny County Health Department Sexually Transmitted Diseases Clinic, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania